CLINICAL TRIAL: NCT05607121
Title: Exogenous Modulation of Visual Perception and Connectivity in Body Dysmorphic Disorder (EMPAC-BDD)
Brief Title: TMS Visual Modulation in Body Dysmorphic Disorder
Acronym: EMPAC-BDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R21MH128815 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-11-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-06

CONDITIONS: Body Dysmorphic Disorders
Keywords: transcranial magnetic stimulation; visual processing; brain connectivity; theta burst stimulation; fMRI
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iTBS then cTBS (Experimental): iTBS day 1, cTBS day 2
  Interventions: Device: intermittent theta burst stimulation; Device: continuous theta burst stimulation
- cTBS then iTBS (Experimental): cTBS day 1, iTBS day 2
  Interventions: Device: intermittent theta burst stimulation; Device: continuous theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — transcranial magnetic stimulation
Device: continuous theta burst stimulation — transcranial magnetic stimulation

SUMMARY:
The goal of this observational study is to test the effects of a type of noninvasive brain stimulation called transcranial magnetic stimulation (TMS) on visual processing in adults with body dysmorphic disorder symptoms when combined with modifying visual attention.

The main goals are to understand, in people with body dysmorphic disorder and people with subclinical body dysmorphic disorder:

* The effects of intermittent and continuous TMS stimulation of parietal brain regions when done right before visual attention modulation on brain functional connections.
* The effects of intermittent and continuous TMS stimulation of parietal brain regions when done right before visual attention modulation on global/holistic visual perception.

Participants will receive one type of TMS (intermittent or continuous) followed immediately by an fMRI brain scan during which they will view images of their faces. On the second day, they will do the same, but receive either the intermittent or continuous TMS stimulation that they did not receive on the first day.

DETAILED DESCRIPTION:
PROJECT SUMMARY

Individuals with body dysmorphic disorder (BDD) misperceive aspects of their appearance to be conspicuously flawed or defective, despite these being unnoticeable or appearing miniscule to others. With convictions of disfigurement and ugliness, they typically have poor insight or delusional beliefs, obsessive thoughts and compulsive behaviors, anxiety, and depression. These result in significant difficulties in functioning, depression, suicide attempts (25%), and psychiatric hospitalization (50%). Despite this, relatively few studies of the neurobiology, and few treatment studies, have been conducted. This underscores a critical need for research to identify novel targets for intervention based on a comprehensive understanding of the pathophysiological mechanisms. Previous research has uncovered mechanisms that may contribute to perceptual distortions, including prominent abnormalities in visual processing systems. These have contributed to a model of diminished global/holistic processing and enhanced local/detailed processing, attributed to "bottom-up" and "top-down" disturbances in perception. Previous experiments using psychophysical tests, novel behavioral visual modulation techniques, and functional magnetic resonance imaging (fMRI) have probed the brain's visual systems responsible for global and local processing and found early evidence that they may be modifiable in BDD. This study will test if further modification could be achieved using noninvasive neuromodulation with repetitive transcranial magnetic stimulation (TMS). Such modulation may be necessary to enhance the effects of behavioral modulation and induce the magnitude of functional changes necessary to achieve clinically meaningful improvements in perceptual experiences in those with BDD. The proposed experiment will determine whether intermittent and continuous TMS enhances and inhibits, respectively, the effects of a behavioral visual modulation strategy on brain connectivity and on global visual processing on a psychophysical task. This will be tested in individuals with clinical BDD and in individuals with subclinical BDD. Results will contribute to a comprehensive mechanistic model of abnormal visual information processing underlying the core symptom domain of misperceptions of appearance. Further, results will be critical for the development and optimization of future combinations of neuromodulation and novel perceptual retraining treatments.

ELIGIBILITY:
Inclusion Criteria:

Body dysmorphic disorder:

Inclusion:

* males or females
* ages 18-40
* meet Diagnostic and Statistical Manual (DSM-5) criteria for Body Dysmorphic Disorder
* have a Body Dysmorphic Disorder version of the Yale-Brown Obsessive-Compulsive Disorder Scale (BDD-YBOCS) score of ≥20
* primary appearance concerns of the face or head area
* medication naïve or medication free for at least 8 weeks prior to enrollment

Subclinical body dysmorphic disorder:

* males or females
* ages 18-40
* have a score on the Dysmorphic Concern Questionnaire of ≥8 (1 standard deviation [STD] above population norms)
* primary appearance concerns of the face or head area
* medication naïve or medication free for at least 8 weeks prior to enrollment

Exclusion Criteria:

Body dysmorphic disorder:

* concurrent major Axis I disorders including substance use disorders, aside from anxiety disorders or depressive disorders as these comorbidities are very common and the sample would otherwise be non-representative; however, BDD must be the primary diagnosis.
* lifetime: bipolar disorder or psychotic disorder
* psychotropic medications, aside from a short half-life sedative/hypnotic for insomnia, or a short half-life benzodiazepine as needed for anxiety but not exceeding a frequency of 3 doses in one week and not to be taken on the days of the training or MRI scan
* current cognitive-behavioral therapy

Subclinical body dysmorphic disorder:

Exclusion:

* meet full DSM-5 criteria for body dysmorphic disorder
* current Axis I disorders including substance use disorders
* lifetime: bipolar disorder or psychotic disorder
* psychotropic medications, aside from a short half-life sedative/hypnotic for insomnia, or a short half-life benzodiazepine as needed for anxiety but not exceeding a frequency of 3 doses in one week and not to be taken on the days of the training or MRI scan
* current cognitive-behavioral therapy

Exclusion criteria for all participants:

* Neurological disorder
* Pregnancy
* Current major medical disorders that may affect cerebral metabolism such as diabetes or thyroid disorders
* Current risk of suicide with a plan and intent
* Ferromagnetic metal implantations or devices (electronic implants or devices, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates)
* Visual acuity worse than 20/35 for each eye as determined by Snellen close vision acuity chart (vision will be tested with corrective lenses if participant uses them).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — We will ask participants to report their identified gender.
Enrollment: 40 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Face inversion effect | Before TMS on Day 2
  In a force-choice recognition task, participants will view sets of upright target faces followed by 2 upright selection faces, and sets of inverted target faces followed by 2 inverted selection faces. They will be instructed to select one of the two faces that is the same as the target face, as quickly and as accurately as possible. The dependent variable is the difference in response times for upright vs. inverted faces.
Face inversion effect | After fMRI on Day 2
  In a force-choice recognition task, participants will view sets of upright target faces followed by 2 upright selection faces, and sets of inverted target faces followed by 2 inverted selection faces. They will be instructed to select one of the two faces that is the same as the target face, as quickly and as accurately as possible. The dependent variable is the difference in response times for upright vs. inverted faces.
Face inversion effect | Before TMS on Day 3
  In a force-choice recognition task, participants will view sets of upright target faces followed by 2 upright selection faces, and sets of inverted target faces followed by 2 inverted selection faces. They will be instructed to select one of the two faces that is the same as the target face, as quickly and as accurately as possible. The dependent variable is the difference in response times for upright vs. inverted faces.
Face inversion effect | After fMRI on Day 3
  In a force-choice recognition task, participants will view sets of upright target faces followed by 2 upright selection faces, and sets of inverted target faces followed by 2 inverted selection faces. They will be instructed to select one of the two faces that is the same as the target face, as quickly and as accurately as possible. The dependent variable is the difference in response times for upright vs. inverted faces.
Body Image States Scale (BISS) | Before fMRI on Day 2
  This scale consists of six items written to assess the following domains of current body experience: (1) dissatisfaction-satisfaction with one's overall physical appearance; (2) dissatisfaction-satisfaction with one's body size and shape; (3) dissatisfaction-satisfaction with one's weight; (4) feelings of physical attractiveness- unattractiveness; (5) current feelings about one's looks relative to how one usually feels; and (6) evaluation of one's appearance relative to how the average person looks.
Body Image States Scale (BISS) | After fMRI on Day 2
  This scale consists of six items written to assess the following domains of current body experience: (1) dissatisfaction-satisfaction with one's overall physical appearance; (2) dissatisfaction-satisfaction with one's body size and shape; (3) dissatisfaction-satisfaction with one's weight; (4) feelings of physical attractiveness- unattractiveness; (5) current feelings about one's looks relative to how one usually feels; and (6) evaluation of one's appearance relative to how the average person looks.
Body Image States Scale (BISS) | Before fMRI on Day 3
  This scale consists of six items written to assess the following domains of current body experience: (1) dissatisfaction-satisfaction with one's overall physical appearance; (2) dissatisfaction-satisfaction with one's body size and shape; (3) dissatisfaction-satisfaction with one's weight; (4) feelings of physical attractiveness- unattractiveness; (5) current feelings about one's looks relative to how one usually feels; and (6) evaluation of one's appearance relative to how the average person looks.
Body Image States Scale (BISS) | After fMRI on Day 3
  This scale consists of six items written to assess the following domains of current body experience: (1) dissatisfaction-satisfaction with one's overall physical appearance; (2) dissatisfaction-satisfaction with one's body size and shape; (3) dissatisfaction-satisfaction with one's weight; (4) feelings of physical attractiveness- unattractiveness; (5) current feelings about one's looks relative to how one usually feels; and (6) evaluation of one's appearance relative to how the average person looks.
Brain connectivity and activation in the dorsal and ventral visual stream while viewing own faces | After TMS on Day 2
  We will obtain fMRI data while participants view photographs of their own face. After preprocessing and analysis we will be able to determine: a) changes in dorsal and ventral visual stream connectivity while naturalistically viewing faces after, compared with before, visual attention modulation. This will be determined for both the fMRI task following iTBS and cTBS. We will also determine, b) associations between changes in brain connectivity with changes in global/local processing (face inversion effect) as a result of iTBS and cTBS.
Brain connectivity and activation in the dorsal and ventral visual stream while viewing own faces | After TMS on Day 3
  We will obtain fMRI data while participants view photographs of their own face. After preprocessing and analysis we will be able to determine: a) changes in dorsal and ventral visual stream connectivity while naturalistically viewing faces after, compared with before, visual attention modulation. This will be determined for both the fMRI task following iTBS and cTBS. We will also determine, b) associations between changes in brain connectivity with changes in global/local processing (face inversion effect) as a result of iTBS and cTBS.
Brain connectivity and activation in the dorsal and ventral visual stream while viewing scrambled faces | After TMS on Day 2
  For an exploratory analysis, we will obtain fMRI data while participants view photographs of scrambled faces, to understand how non-face related visual processing is affected by TMS. After preprocessing and analysis we will be able to determine: a) changes in dorsal and ventral visual stream connectivity while naturalistically viewing faces after, compared with before, visual attention modulation. This will be determined for both the fMRI task following iTBS and cTBS. We will also determine, b) associations between changes in brain connectivity with changes in global/local processing (face inversion effect) as a result of iTBS and cTBS.
Brain connectivity and activation in the dorsal and ventral visual stream while viewing scrambled faces | After TMS on Day 3
  For an exploratory analysis, we will obtain fMRI data while participants view photographs of scrambled faces, to understand how non-face related visual processing is affected by TMS. After preprocessing and analysis we will be able to determine: a) changes in dorsal and ventral visual stream connectivity while naturalistically viewing faces after, compared with before, visual attention modulation. This will be determined for both the fMRI task following iTBS and cTBS. We will also determine, b) associations between changes in brain connectivity with changes in global/local processing (face inversion effect) as a result of iTBS and cTBS.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Feusner, M.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Wong WW, Rangaprakash D, Larson MS, Diaz-Fong JP, Tadayonnejad R, Leuchter AF, Feusner JD. Can excitatory neuromodulation change distorted perception of one's appearance? Brain Stimul. 2021 Sep-Oct;14(5):1197-1200. doi: 10.1016/j.brs.2021.07.010. Epub 2021 Jul 30. No abstract available. PMID 34339891
- See also: Published manuscript of the pilot study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9007239/